CLINICAL TRIAL: NCT01831336
Title: BIOTRONIK - SaFety and Performance Registry for an All-comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice - III Belgium
Brief Title: BIOFLOW-III Belgium Satellite Registry
Status: Completed | Type: Observational
Sponsor: Biotronik Belgium NV (Industry)
Responsible Party: Sponsor
Other Study IDs: G1215
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: International; Multicenter; Observational registry; Orsiro Drug Eluting Stent (DES); Stenting; Treatment of Coronary Artery Disease; Coronary revascularization; Percutaneous Coronary Intervention; STEMI; NSTEMI; Ischemia; Angina; Subgroups; Acute Myocardial Infarction; Diabetes; Small Vessels; Chronic Total Occlusion (CTO)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro DES

SUMMARY:
This registry is a clinical post-market evaluation of the Orsiro LESS in subjects requiring coronary revascularization with Drug Eluting Stents (DES).

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD), treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedural success. However, the medium to long-term complications range from rather immediate elastic recoil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30%-50%. Such rates of recurrence have serious economic consequences.

Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in de novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20%-40% of cases, necessitating repeat procedures.

The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilised on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in a better safety profile as compared to BMS with systemic drug administration.

These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease. This observational registry is designed to investigate and collect clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in an all-comers patient population in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease
* Subject has signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow-up assessments
* Subject is ≥ 18 years

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Pregnancy
* Known intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not reached yet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers patient population with all subjects requiring coronary revascularization with a Drug Eluting Stent (DES)
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non-Q wave Myocardial Infarction (MI), Emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Target Vessel Revascularization (TVR) | 6 and 12 months
  Any repeat revascularization of the target vessel.
Target Lesion Revascularization (TLR) | 6 and 12 months
  Any repeat revascularization of the target lesion.
Stent Thrombosis | 6 and 12 months
  Definite, Probable and Possible Stent Thrombosis
Clinical Device Success | At time of intervention
  Successful delivery and deployment of the investigational stent(s) at the intended target lesion (this includes successful delivery and deployment of multiple overlapping stents) and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without use of a device outside the assigned treatment strategy. Standard predilation catheters and post-dilation catheters (if applicable) may be used.
Clinical Procedural Success | During the hospital stay to a maximum of the first seven days post index procedure
  Successful delivery and deployment of the investigational stent(s) at the intended target lesion (this includes successful delivery and deployment of multiple overlapping stents, if applicable) and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% of the target lesion as observed by visual estimate without using any adjunctive device* without the occurrence of ischemia-driven major adverse cardiac event (ID-MACE) during the hospital stay to a maximum of the first seven days post index procedure.
Target Lesion Failure (TLF) | 6 months
  Composite of cardiac death, target vessel Q-wave or non-Q wave Myocardial Infarction (MI), Emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Legrand, Prof. Dr., Principal Investigator — CHU Liege (Hospitalo-Facultaire Universitaire de Liège)
Locations (8):
- Belgium (8):
  - UCL St. Luc, Brussels
  - Brussels Heart Center, Brussels
  - CHU Charleroi, Charleroi
  - Grand Hopital de Charleroi Saint Joseph, Gilly
  - CHR de la Citadelle, Liège
  - CHU Liège, Liège
  - Brussels Heart Center St Pierre, Ottignies
  - UCL de Mont Godine, Yvoir